CLINICAL TRIAL: NCT05028010
Title: Enhancing the Health Extension Workers Capacity for Promotion of Maternal and Child Nutrition in Northwest Ethiopia: Applying the Pender's Health Promotion Model
Brief Title: Enhancing the Health Extension Workers Capacity for Promotion of Maternal and Child
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Gondar (Other)
Collaborators: International Institute for Primary Health Care-Ethiopia (IIfPHC-E) (Unknown)
Responsible Party: Principal Investigator, Wubet Worku Takele, Mr., University of Gondar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V/P/RCS/05/837/21
Record Dates: First submitted 2021-08-09; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Behavior Problem
Keywords: Community health workers; Maternal and Child nutrition
MeSH Terms: conditions — Mental Disorders | interventions — Capacity Building

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study aimed to look at the impact of model-based education on the improvement of nutrition promotion.
Masking Description: No masking will be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental): There will be one arm, intervention group.
  Interventions: Behavioral: Capacity building

INTERVENTIONS:
Behavioral: Capacity building — Four days of training on the promotion of maternal and child nutrition will be given. The training will be based on Pender's health promotion model. Supportive supervision will be conducted.

SUMMARY:
Background: Maternal and child nutrition is a lingering public health concern, affecting the lives of the most vulnerable individuals, in particular mothers and children. To counteract the burden, the Ethiopian government has applied various strategies, including incorporating the promotion of nutrition as one package of primary health care provided by the health extension workers (HEWs). However, the provider's knowledge, promotion skill, and competency for promoting maternal and child nutrition have not been examined. Moreover, health extension workers have been promoting using the traditional model of education and indicating the need for continuous professional development to strengthen the workforce. Thus, the study is aimed to assess and enhance the health extension worker's capacity in promoting maternal and child nutrition through comprehensive and evidence-based capacity-building training.

Methods: A quasi-experimental study will be employed among 92 health extension workers. A baseline study, involving both qualitative and quantitative studies will be conducted to identify the gaps in maternal and child nutrition promotion. The knowledge, promotion as well as counseling skills of the HEWs will be assessed using a self-administered questionnaire and observational checklist, respectively. The intervention will involve training, supportive supervision, and coaching in a real environment. A four-day training will be given, which will be followed by supportive supervision of expert supervisors. Further, the greet, ask, listen, identify, discuss, recommend, and agree counseling model with Pender's health promotion model will be applied to enhance HEWs promotion skill. A post-test aimed at assessing the knowledge and counseling competency will be conducted and the pretest and posttest results will be compared using a t-test. Factors affecting both knowledge and counseling capacity will be assessed using binary logistic and linear regression, respectively. Similarly, a qualitative study will be used to explore promotion skills.

Discussion: Given there are problems associated with the knowledge and counseling skills of HEWs in Ethiopia, nutrition education using a well-designed and comprehensive strategy would bring a positive impact on professionals' promotion capacity thereby improving mothers/caregivers' behavior regarding child and maternal nutrition. The evidence will also enforce nutrition programmers and the Amhara regional health bureau to end maternal and child undernutrition.

ELIGIBILITY:
Inclusion Criteria:

-All health extension workers working in the study area will be included.

Exclusion Criteria:

* Not any

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changed the knowledge of community health workers about maternal and child nutrition | Four weeks
  They will be expected to be knowledgeable about maternal and child nutrition. It will be measured using self-administer questionnaire.
Changed the community health workers counseling capacity. | Four weeks
  The professionals counseling skill is expected to be improved through the training. This outcome will be measured using observational checklist. Participants will be expected to counsel pregnant women, children on breastfeeding and complementary feeding, and data collectors will fill out the checklist accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Gondar Zone, Gonder, Ethiopia

IPD SHARING:
Plan to Share IPD: No